CLINICAL TRIAL: NCT05752916
Title: Intravenous Thrombolysis With Recombinant Human TNK Tissue-type Plasminogen Activator (rhTNK-tPA) for Acute Non-large Vessel Occlusion in Extended Time Window--A Multicenter, Prospective, Randomized, Open-label, Blinded End-point Trial
Brief Title: Intravenous Thrombolysis With rhTNK-tPA for Acute Non-large Vessel Occlusion in Extended Time Window
Acronym: OPTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: CSPC Mingfule Pharmaceutical (Guangzhou) Co., Ltd. (Industry); Beijing Hospitals Authority (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: [2022]205
Record Dates: First submitted 2023-02-09; First posted 2023-03-03 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-04

CONDITIONS: Acute Ischemic Stroke
Keywords: acute ischemic stroke; extended time window; non-large vessel occlusion; intravenous thrombolysis
MeSH Terms: conditions — Ischemic Stroke | interventions — Platelet Aggregation Inhibitors; Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: prospective, randomized, open label, blinded-endpoint (PROBE)
Who Masked: Outcomes Assessor
Masking Description: An imaging core laboratory (ICL) is to provide an unbiased assessment of imaging measures. They are knowledgeable in the analysis of neuroradiological images and will be blinded, i.e. unaware of the patient's treatment allocation and trial outcome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intravenous rhTNK-tPA (Experimental): rhTNK-tPA(0.25mg/kg) given as a single, intravenous bolus immediately upon randomization. Experimental treatment will be administered as a single intravenous bolus over 5-10 seconds as per the standard manufacturers' instructions for use.
  Interventions: Drug: rhTNK-tPA
- Standard Medical Treatment (Active Comparator): Antiplatelet therapy (aspirin or clopidogrel alone) at the discretion of local investigators according to Chinese Guidelines for Diagnosis and Treatment of Acute Ischemic Stroke 2023.
  Interventions: Drug: Antiplatelet Agents

INTERVENTIONS:
Drug: rhTNK-tPA — Recombinant human TNK tissue-type plasminogen activator. Patients will receive intravenous rhTNK-tPA (0.25mg/kg, maximum 25mg, administered as a bolus over 5-10 seconds).
  Arms: Intravenous rhTNK-tPA
Drug: Antiplatelet Agents — Aspirin (150-300mg) is offered to patients allocated in the control arm, unless contraindicated. According to Chinese Guidelines for Diagnosis and Treatment of Acute Ischemic Stroke 2023, 150-300mg aspirin alone is recommended for acute stroke treatment in patients who are otherwise eligible for intravenous thrombolysis or EVT as soon as possible (Class 1 of recommendation, Level A of evidence). The aspirin dose can be changed to 50-300 mg/day after the acute phase. Clopidogrel is indicated as an alternative in case of aspirin intolerance (Class 2 of recommendation, Level C of evidence)
  Other Names: Aspirin; Clopidogrel
  Arms: Standard Medical Treatment

SUMMARY:
This study is designed to evaluate the efficacy of IV rhTNK-tPA between 4.5 to 24 hours from symptom onset in patients presenting with a non-large vessel occlusion ischemic stroke.

DETAILED DESCRIPTION:
OPTION is a multicenter, prospective, randomized, open-label, blinded end-point (PROBE) controlled trial of thrombolysis with rhTNK-tPA versus standard of care. A total of 568 patients will be enrolled at approximately 40 centers around China.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute ischemic stroke
* Age≥18 years
* Pre-stroke mRS score≤1 points
* Disabling stroke defined as follows:

  * Baseline NIHSS score 6-25 at the time of randomization,
  * Or NIHSS 4-5 with disabling deficit (e.g. hemianopia, aphasia, loss of hand function) as determined by the managing clinician
* Onset (last-seen-well) time to treatment time between 4.5 and 24 hours
* Written informed consent from patients or legally responsible representatives
* The presence of a Target Mismatch on CT perfusion: ischemic core volume<50ml (defined as rCBF<30%), mismatch ratio≥1.2 (Tmax>6 sec lesion/core volume lesion), mismatch volume≥10ml

Exclusion Criteria:

* Treatment with a thrombolytic within the last 72 hours or intention to receive intravenous thrombolysis
* Contraindication to thrombolysis
* Planned or anticipated treatment with endovascular therapy
* Rapidly improving symptoms, particularly if in the judgment of the managing clinician that the improvement is likely to result in a NIHSS score<4 at randomization
* Pregnancy or lactating; formal testing needed in women of childbearing potential
* Brain tumor (with mass effect)
* Hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
* Impairment in coagulation due to comorbid disease or anticoagulant use. If on warfarin, international normalized ratio (INR) >1.7 or prothrombin time >15s; if use of any direct oral anticoagulant within the last 48 hours; if use of heparin/heparinoid within the last 24 hours
* Use of glycoprotein Ⅱb-Ⅲa inhibitors within the last 72 hours
* Baseline platelet count <100,000/μL
* Undergoing hemodialysis or peritoneal dialysis; known severe renal insufficiency with glomerular filtration rate <30ml/min or serum creatinine >220mmol/L (2.5mg/dl)
* Suspected aortic dissection
* Major surgery or biopsy within the last 1 month
* Any active bleeding within the previous 1 month (including gastrointestinal or urinary bleeding)
* Known severe, life-threatening allergy (more severe than skin rash) to contrast agents
* Severe, uncontrolled hypertension (systolic blood pressure >185mmHg or diastolic blood pressure >110mmHg)
* Any terminal illness such that the patient would not be expected to survive more than half a year
* Current participation in any investigational study that may confound outcome assessment of the study
* Any condition that, in the judgement of the investigator, is inappropriate for participation in the trial or could impose hazards to the patient (e.g. inability to understand and/or follow the study procedures and/or follow-up due to mental disorders, cognitive or emotional disorders)

Specific Neuroimaging Exclusion Criteria:

* Evidence of acute intracranial hemorrhage
* Acute large vessel occlusion on magnetic resonance/ computed tomography angiography, including internal carotid artery (ICA), middle cerebral artery M1 segment (MCA-M1）, vertebral artery and basilar artery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Excellent functional outcome | 90±7 days
  Proportion of subjects with mRS 0-1 at 90±7 days

SECONDARY OUTCOMES:
modified Rankin Scale (mRS) score | 90±7 days
  Ordinal distribution of mRS at 90±7 days; modified Rankin scale (range, 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death)
Good functional outcome | 90±7 days
  Proportion of subjects with mRS 0-2 at 90±7 days
Rate of successful reperfusion | 24 hours (-2/+12 hours)
  >90% reduction of the Tmax>6s lesion volumes between the baseline and early follow-up at 24 hours (-2/+12 hours)
Infarct volume at 24 hours (-2/+12 hours) | 24 hours (-2/+12 hours)
  The infarct volume is determined on evaluated on NCCT at 24 hours (-2/+12 hours)
Early clinical recovery | 24 hours (-2/+12 hours)
  Proportion of subjects with NIHSS score≥8 improved compared with baseline or with NIHSS 0-1 at 24 hours (-2/+12 hours)
Change of National Institutes of Health Stroke Scale (NIHSS) | 7±2 days
  Change of NIHSS score from baseline to 7 days (±2days)
Functional health status and quality of life | 90±7 days
  Functional health status and quality of life (EQ-5D-5L) at 90±7 days

OTHER OUTCOMES:
Incidence of clinically significant intracranial hemorrhage | 36 hours
  Incidence of sICH (Heidelberg criteria) measured at 36 hours
Incidence of major bleeding | 90±7 days
  Incidence of major bleeding defined as GUSTO severe/life threatening or moderate bleeds measured at 90±7 days
All-cause mortality | 90±7 days
  All-cause mortality at 90±7 days

CONTACTS AND LOCATIONS:
Overall Officials: Junwei Hao, MD, Principal Investigator — Xuanwu Hospital, Beijing; Qingfeng Ma, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma G, Mo R, Zuo Y, Ma Q, Zhao G, Yao X, Liang J, Zhou L, He Y, Long F, Yuan Z, Liu L, Han G, Tan Y, Ai Z, Cai C, Liu J, Zhang L, Yang H, Yi T, Li L, Fu Y, Zhang Y, Shao X, Yu Z, Wu S, Du Y, Mao L, Guo H, Chen X, Chen Y, Zhao Q, Chi L, Liu Y, Zhang H, Li G, Meng S, Wu Y, Wu J, Jiang Z, Lei S, Gao D, Zhong L, Fiehler J, Wang D, Nguyen TN, Saver JL, Hao J; OPTION Investigators. Tenecteplase for Acute Non-Large Vessel Occlusion 4.5 to 24 Hours After Ischemic Stroke: The OPTION Randomized Clinical Trial. JAMA. 2026 Feb 5:e260210. doi: 10.1001/jama.2026.0210. Online ahead of print. PMID 41642827